CLINICAL TRIAL: NCT03390478
Title: MIND&GAIT - Promoting Independent Living in Frail Older Adults by Improving Cognition and Gait Ability and Using Assistive Products
Brief Title: Promoting Independent Living in Frail Older Adults by Improving Cognition and Gait Ability and Using Assistive Products
Acronym: MIND&GAIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Enfermagem de Coimbra (Other)
Collaborators: Instituto Politécnico de Coimbra (Unknown); Instituto Politécnico de Leiria (Other); Polytechnic University of Santarém (Other)
Responsible Party: Principal Investigator, Joao Apostolo, João Luís Alves Apóstolo, Escola Superior de Enfermagem de Coimbra
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CT_MIND&GAIT
Record Dates: First submitted 2017-12-29; First posted 2018-01-04 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Frailty; Cognition; Mild Cognitive Impairment
Keywords: Frailty; Aged; Cognitive Stimulation; Technology
MeSH Terms: conditions — Frailty; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Participants will be assigned in two groups, a control group who will receive institutional usual care and an experimental group who will receive the combined intervention.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The randomization process it will be done in https://www.random.org/ by an independent person.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The participants that will be assign to the control group will receive institutional usual care.
- Combined Intervention Group (Experimental): The participants that will be assigned to the experimental group will receive the Combined Intervention Program
  Interventions: Other: Combined Intervention Group

INTERVENTIONS:
Other: Combined Intervention Group — Experimental: Combined Intervention Program is composed by a Cognitive Stimulation Program (CSP), a Physical Activity Program (PAP) and Animal Assisted Therapy (AAT). During the PAP participants that use rolling-walkers, will do PAP using the Auto-Blocking kit mechanism for rolling walkers (ABMRW).
  Arms: Combined Intervention Group

SUMMARY:
A strategy involving 6 partners was planned, targeting the components of education, innovation, and practice-based research with knowledge transfer into clinical practice.The project MIND&GAIT aims to promote independent living in frail older people through the development of innovative initiatives and systems to improve cognition and gait ability. A structured and integrated Combined Intervention (CI) will be developed, composed by: cognitive stimulation program, an animal-assisted therapy program, a physical activity program. Moreover, an auto-blocking mechanism for rolling walkers will be developed and implemented in this study. The results of the study and all the material that was used, will be disseminated in a web platform.

DETAILED DESCRIPTION:
In this growing context of aging societies, the number of institutionalized older adults tends to increase. Several reasons lead to the institutionalization of older people, including physical and cognitive decline. In Portugal,in the population aged over 60 years, there was approximately 160,287 people with dementia, which corresponds to 5.91% of the people covered by these age groups. Mild cognitive impairment (MCI) is considered as an intermediate state between normal cognitive ageing and mild dementia, particularly in older people. It is increasingly recognized as a major health problem associated with an increased risk for dementia. Cognitive health maintenance is essential for preventing cognitive impairment and delaying the onset of dementia, dependency, and (in)ability to self-care. In older people with cognitive decline, cognitive stimulation can be a promising intervention for reducing depressive symptoms and depressive vulnerability, improving their quality of life. On the other hand, healthy ageing has traditionally focused on disease prevention, but greater efforts are needed to reduce frailty and dependency, and maintain independent physical and cognitive function among older adults. The aging process associated with a sedentary lifestyle can lead to the decline of some physical capacities. Maintaining functional status and reducing age-related morbidity is an important part of active ageing policies; it promotes independent living, improves the quality of life, and reduces health care costs. In this way exercise programs reduce age-related decline in functional capacity and maintain muscle strength and mass among adults aged 65-85 years.

The research team intend to intervene in the promotion of active ageing, including physical exercise and activities that promote the delay and/or maintenance of the cognitive and physical health of frail older people.

In this way, a randomized controlled trial will be conducted by the research team, composed by two arms: experimental group (CI group) and control group. The aim of this study is to assess the impact of the CI program on frail older people. The evaluation of the effectiveness of the Combined Intervention will have the following methodology:

- Sample Test: For sample size calculation it was used the software G*Power 3.1.9.2. Power analysis was based on a type I error of 0.05; power of 0.80; effect size f=0.30; and ANOVA: repeated measures between factors determined a total sample size of 62.Participants with more than 65 or more years will be recruited from two homes for the aged. Participants will be randomly distributed in groups of 8, in the control group and in the experimental group. Participants will be classified as having mild to moderate cognitive decline and risk of fall from mild to moderate. The control group will receive usual care.

-Intervention: The combined intervention will be implemented over 21 weeks, 4 times a week. Cognitive Stimulation Program (CSP) will be applied once a week and Physical Activity Program (PAP) 3 times a week for 30-60 min. Participants using rolling walkers will benefit from the autoblocking kit mechanism for rolling walkers mechanism (ABMRW) during the execution of the PAP.

-Data analysis: Statistical analysis will be performed through repeated meaures and ANOVA. Age, gender, and initial scores of depression and Activities of Daily Living (ADLs) will be introduced as covariates. Intention-to-treat analysis will be done to analyze the data of the people who left the study.

ELIGIBILITY:
Inclusion Criteria:

* Older adults, age 65 or above;
* Older adults with the ability to consent in an informed manner their participation in the study;
* Older adults with clinical conditions that allow them to participate in the combined intervention;
* Older adults with mild to moderate cognitive frailty criteria as per the 6-CIT scale;
* Older adults with mild to moderate depressive status as per the Geriatric Depression Scale (15 items version).
* Older adults that present mild to moderate risk of fall tracked by Tinetti Index;
* Older adults with physical frailty tracked by the biomechanical gait parameters.

Exclusion Criteria:

* Older adults without a stable clinical condition;
* Older adults with a cardiac condition that enables them practice of physical activity;
* Older adults that do not have the desire of participate in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2018-05-23 (Actual); Study Completion 2018-10-22 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the participant's Cognition | Intermediate assessment (week 12)
  Outcome measure: "Montreal Cognitive Assessment (MoCA)" - Portuguese version of Freitas, S., Simões, M. R., Santana, I., Martins, C. & Nasreddine, Z. (2013).
Change from Baseline in the participant's Cognition | Post-intervention assessment (week 21)
  Outcome measure: "Montreal Cognitive Assessment (MoCA)" - Portuguese version of Freitas, S., Simões, M. R., Santana, I., Martins, C. & Nasreddine, Z. (2013).
Change from Baseline in the participant's Physical Frailty | Intermediate assessment (week 12)
  Outcome measure: "Gait B" with a stopwatch that will be adapted to the specific context. It will also be measure biomechanical parameters of gait using the Novel EMED-X pressure platform. The fall risk it will be measure with "Tinetti Index", original version of Tinetti, Wiliams and Mayewski (1986), translated and adapted to portuguese by Elisa Petiz (2001).
Change from Baseline in the participant's Physical Frailty | Post-intervention assessment (week 21)
  Outcome measure: "Gait B" with a stopwatch that will be adapted to the specific context. It will also be measure biomechanical parameters of gait using the Novel EMED-X pressure platform. The fall risk it will be measure with "Tinetti Index", original version of Tinetti, Wiliams and Mayewski (1986), translated and adapted to portuguese by Elisa Petiz (2001).

SECONDARY OUTCOMES:
Change from Baseline in the participant's Activities of Daily Living | Intermediate assessment (week 12)
  Outcome measure: "Barthel ADL Index - Portuguese version"
Change from Baseline in the participant's Activities of Daily Living | Post-intervention assessment (week 21)
  Outcome measure: "Barthel ADL Index - Portuguese version"

CONTACTS AND LOCATIONS:
Overall Officials: João Apóstolo, Aggregation, Principal Investigator — Nursing School of Coimbra (ESEnfC)
Locations (1):
- Health Sciences Research Unit: Nursing, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bradley SM, Hernandez CR. Geriatric assistive devices. Am Fam Physician. 2011 Aug 15;84(4):405-11. PMID 21842786
- [Background] Peretz C, Korczyn AD, Shatil E, Aharonson V, Birnboim S, Giladi N. Computer-based, personalized cognitive training versus classical computer games: a randomized double-blind prospective trial of cognitive stimulation. Neuroepidemiology. 2011;36(2):91-9. doi: 10.1159/000323950. Epub 2011 Feb 10. PMID 21311196
- [Background] Tinetti ME, Williams TF, Mayewski R. Fall risk index for elderly patients based on number of chronic disabilities. Am J Med. 1986 Mar;80(3):429-34. doi: 10.1016/0002-9343(86)90717-5. PMID 3953620
- [Background] Reeves ND, Narici MV, Maganaris CN. Musculoskeletal adaptations to resistance training in old age. Man Ther. 2006 Aug;11(3):192-6. doi: 10.1016/j.math.2006.04.004. Epub 2006 Jun 19. PMID 16782393
- [Background] Skelton DA, Beyer N. Exercise and injury prevention in older people. Scand J Med Sci Sports. 2003 Feb;13(1):77-85. doi: 10.1034/j.1600-0838.2003.00300.x. PMID 12535321
- [Background] Narici MV, Maganaris CN, Reeves ND, Capodaglio P. Effect of aging on human muscle architecture. J Appl Physiol (1985). 2003 Dec;95(6):2229-34. doi: 10.1152/japplphysiol.00433.2003. Epub 2003 Jul 3. PMID 12844499
- [Background] Narici MV, Maffulli N. Sarcopenia: characteristics, mechanisms and functional significance. Br Med Bull. 2010;95:139-59. doi: 10.1093/bmb/ldq008. Epub 2010 Mar 2. PMID 20200012
- [Background] Macaluso A, De Vito G. Muscle strength, power and adaptations to resistance training in older people. Eur J Appl Physiol. 2004 Apr;91(4):450-72. doi: 10.1007/s00421-003-0991-3. Epub 2003 Nov 25. PMID 14639481
- [Background] Puthoff ML, Nielsen DH. Relationships among impairments in lower-extremity strength and power, functional limitations, and disability in older adults. Phys Ther. 2007 Oct;87(10):1334-47. doi: 10.2522/ptj.20060176. Epub 2007 Aug 7. PMID 17684086
- [Background] Skelton DA. Effects of physical activity on postural stability. Age Ageing. 2001 Nov;30 Suppl 4:33-9. doi: 10.1093/ageing/30.suppl_4.33. No abstract available. PMID 11769787
- [Background] Paiva, Diana S; Apóstolo, João L. A. 2015. Estudo de adaptação transcultural e validação do Six Item Cognitive Impairment Test . In J. Apóstolo & M. Almeida (Eds). Elderly Health Care Nursing. Monographic Series - Health Sciences Education and Research, 3 - 18. ISBN: 978-989-99426-1-5. Coimbra: Unidade de Investigação em Ciências da Saúde: Enfermagem (UICISA: E) ESEnfC.
- [Background] Guideline for the prevention of falls in older persons. American Geriatrics Society, British Geriatrics Society, and American Academy of Orthopaedic Surgeons Panel on Falls Prevention. J Am Geriatr Soc. 2001 May;49(5):664-72. No abstract available. PMID 11380764
- [Background] Carter ND, Kannus P, Khan KM. Exercise in the prevention of falls in older people: a systematic literature review examining the rationale and the evidence. Sports Med. 2001;31(6):427-38. doi: 10.2165/00007256-200131060-00003. PMID 11394562
- [Background] Bandeira, M. L., Azevedo, A. B., Gomes, C. S., Tomé, L. P., Mendes, M. F., Baptista, M. I., & Moreira, M. J. (2014). Dinâmicas demográficas e envelhecimento da população portuguesa( 1950-2011): evolução e perspetivas. Lisboa: Francisco Manuel dos Santos.
- [Background] Santana I, Farinha F, Freitas S, Rodrigues V, Carvalho A. [The Epidemiology of Dementia and Alzheimer Disease in Portugal: Estimations of Prevalence and Treatment-Costs]. Acta Med Port. 2015 Mar-Apr;28(2):182-8. Epub 2015 May 29. Portuguese. PMID 26061508
- [Background] Sousa, R. (2015). Prevenção de quedas na população geriátrica artigo de revisão. Coimbra, Portugal: Faculdade de Medicina da Universidade de Coimbra.
- [Background] Bauman A, Merom D, Bull FC, Buchner DM, Fiatarone Singh MA. Updating the Evidence for Physical Activity: Summative Reviews of the Epidemiological Evidence, Prevalence, and Interventions to Promote "Active Aging". Gerontologist. 2016 Apr;56 Suppl 2:S268-80. doi: 10.1093/geront/gnw031. PMID 26994266
- [Background] American College of Sports Medicine; Chodzko-Zajko WJ, Proctor DN, Fiatarone Singh MA, Minson CT, Nigg CR, Salem GJ, Skinner JS. American College of Sports Medicine position stand. Exercise and physical activity for older adults. Med Sci Sports Exerc. 2009 Jul;41(7):1510-30. doi: 10.1249/MSS.0b013e3181a0c95c. PMID 19516148
- [Background] Nelson ME, Rejeski WJ, Blair SN, Duncan PW, Judge JO, King AC, Macera CA, Castaneda-Sceppa C; American College of Sports Medicine; American Heart Association. Physical activity and public health in older adults: recommendation from the American College of Sports Medicine and the American Heart Association. Circulation. 2007 Aug 28;116(9):1094-105. doi: 10.1161/CIRCULATIONAHA.107.185650. Epub 2007 Aug 1. PMID 17671236
- [Background] Paterson DH, Warburton DE. Physical activity and functional limitations in older adults: a systematic review related to Canada's Physical Activity Guidelines. Int J Behav Nutr Phys Act. 2010 May 11;7:38. doi: 10.1186/1479-5868-7-38. PMID 20459782
- [Background] Tak E, Kuiper R, Chorus A, Hopman-Rock M. Prevention of onset and progression of basic ADL disability by physical activity in community dwelling older adults: a meta-analysis. Ageing Res Rev. 2013 Jan;12(1):329-38. doi: 10.1016/j.arr.2012.10.001. Epub 2012 Oct 10. PMID 23063488
- [Background] European Union. (2013). Action Group A3 on Prevention and early diagnosis of frailty and functional decline, both physically and cognitive, in older people: A compilation of good practices. The European Innovation Partnership on Active and Healthy Ageing.
- [Background] Apostolo J, Cooke R, Bobrowicz-Campos E, Santana S, Marcucci M, Cano A, Vollenbroek M, Holland C. Effectiveness of the interventions in preventing the progression of pre-frailty and frailty in older adults: a systematic review protocol. JBI Database System Rev Implement Rep. 2016 Jan;14(1):4-19. doi: 10.11124/jbisrir-2016-2467. No abstract available. PMID 26878916
- [Background] Apostolo J, Cooke R, Bobrowicz-Campos E, Santana S, Marcucci M, Cano A, Vollenbroek-Hutten M, Germini F, Holland C. Predicting risk and outcomes for frail older adults: an umbrella review of frailty screening tools. JBI Database System Rev Implement Rep. 2017 Apr;15(4):1154-1208. doi: 10.11124/JBISRIR-2016-003018. PMID 28398987
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Kojima G. Prevalence of Frailty in Nursing Homes: A Systematic Review and Meta-Analysis. J Am Med Dir Assoc. 2015 Nov 1;16(11):940-5. doi: 10.1016/j.jamda.2015.06.025. Epub 2015 Aug 6. PMID 26255709
- [Background] Sternberg SA, Wershof Schwartz A, Karunananthan S, Bergman H, Mark Clarfield A. The identification of frailty: a systematic literature review. J Am Geriatr Soc. 2011 Nov;59(11):2129-38. doi: 10.1111/j.1532-5415.2011.03597.x. Epub 2011 Sep 21. PMID 22091630
- [Background] Langlois F, Vu TT, Kergoat MJ, Chasse K, Dupuis G, Bherer L. The multiple dimensions of frailty: physical capacity, cognition, and quality of life. Int Psychogeriatr. 2012 Sep;24(9):1429-36. doi: 10.1017/S1041610212000634. Epub 2012 Apr 25. PMID 22717010
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Varadhan R, Seplaki CL, Xue QL, Bandeen-Roche K, Fried LP. Stimulus-response paradigm for characterizing the loss of resilience in homeostatic regulation associated with frailty. Mech Ageing Dev. 2008 Nov;129(11):666-70. doi: 10.1016/j.mad.2008.09.013. Epub 2008 Sep 30. PMID 18938195
- [Background] Clegg A, Young J, Iliffe S, Rikkert MO, Rockwood K. Frailty in elderly people. Lancet. 2013 Mar 2;381(9868):752-62. doi: 10.1016/S0140-6736(12)62167-9. Epub 2013 Feb 8. PMID 23395245
- [Background] Fried LP, Ferrucci L, Darer J, Williamson JD, Anderson G. Untangling the concepts of disability, frailty, and comorbidity: implications for improved targeting and care. J Gerontol A Biol Sci Med Sci. 2004 Mar;59(3):255-63. doi: 10.1093/gerona/59.3.m255. PMID 15031310
- [Background] Elliott, S. M. (2015). The Psychological Benefits of Animal Assisted Therapy on Elderly Nursing Home Patients. University of Akron: Ohio?s Polytechnic University.
- [Background] Bono, A. V., BenVenuti, C., Buzzi, M., CiAtti, R., ChiARelli, V., ChiAMBRetto, P., ... & PinCiRoli, M. (2015). Effects of animal assisted therapy (AAT) carried out with dogs on the evolution of mild cognitive impairment. G Gerontol, 63, 32-36.
- [Background] Aguirre E, Hoare Z, Spector A, Woods RT, Orrell M. The effects of a Cognitive Stimulation Therapy [CST] programme for people with dementia on family caregivers' health. BMC Geriatr. 2014 Mar 14;14:31. doi: 10.1186/1471-2318-14-31. PMID 24628705
- [Background] Yuill N, Hollis V. A systematic review of cognitive stimulation therapy for older adults with mild to moderate dementia: an occupational therapy perspective. Occup Ther Int. 2011 Dec;18(4):163-86. doi: 10.1002/oti.315. Epub 2011 Mar 21. PMID 21425381
- [Background] Apóstolo, J., & Cardoso, D. (2014a). Estimulação Cognitiva em Idosos - Síntese da Evidência e Intervenção. In L. coord. Loureiro (Ed.), Literacia em Saúde Mental - Capacitar as pessoas e as Comunidades para Agir (pp. 157?183). Coimbra: Unidade de Investigação em Ciências da Saúde: Enfermagem e Escola Superior de Enfermagem de Coimbra.
- [Background] Apóstolo, J., & Cardoso, D. (2014b). Estimulação Cognitiva em Idosos - Síntese da Evidência e Intervenção: Programa de Manutenção. In M. Apóstolo, J.; Almeida (Ed.), Envelhecimento, Saúde e Cidadania 2: Monographic Series Health Sciences Education and Research (pp. 37?66). Coimbra.
- [Background] Cognitive stimulation and brain fitness. In Action Group A3 on Prevention and early diagnosis of frailty and functional decline, both physically and cognitive, in older people: A compilation of good practices. The European Innovation Partnership on Active and Healthy Ageing.
- [Background] Apostolo JL, Cardoso DF, Rosa AI, Paul C. The effect of cognitive stimulation on nursing home elders: a randomized controlled trial. J Nurs Scholarsh. 2014 May;46(3):157-66. doi: 10.1111/jnu.12072. Epub 2014 Mar 5. PMID 24597922
- [Background] Apostolo J, Holland C, O'Connell MD, Feeney J, Tabares-Seisdedos R, Tadros G, Campos E, Santos N, Robertson DA, Marcucci M, Varela-Nieto I, Crespo-Facorro B, Vieta E, Navarro-Pardo E, Selva-Vera G, Balanza-Martinez V, Cano A. Mild cognitive decline. A position statement of the Cognitive Decline Group of the European Innovation Partnership for Active and Healthy Ageing (EIPAHA). Maturitas. 2016 Jan;83:83-93. doi: 10.1016/j.maturitas.2015.10.008. Epub 2015 Oct 22. PMID 26520249
- [Background] Apóstolo, J., Loureiro, L., Reis, I., Silva, I., Cardoso, D., & Sfectcu, R. (2014). Contribuição para a adaptação da Geriatric Depression Scale -15 para a língua portuguesa. Revista de Enfermagem Referência, Série 3 (3), 65?73.
- [Background] American College of Sports Medicine. (2013). ACSM's guidelines for exercise testing and prescription. Lippincott Williams & Wilkins. ISBN-13: 978-1609136055.
- [Background] Ramalho F, Carnide F, Santos-Rocha R, Andre HI, Moniz-Pereira V, Machado ML, Veloso AP. Community-Based Exercise Intervention for Gait and Functional Fitness Improvement in an Older Population: Study Protocol. J Aging Phys Act. 2017 Jan;25(1):84-93. doi: 10.1123/japa.2015-0290. Epub 2016 Sep 6. PMID 27623478
- [Background] Schwenk M, Howe C, Saleh A, Mohler J, Grewal G, Armstrong D, Najafi B. Frailty and technology: a systematic review of gait analysis in those with frailty. Gerontology. 2014;60(1):79-89. doi: 10.1159/000354211. Epub 2013 Aug 15. PMID 23949441
- [Background] Van Abbema R, De Greef M, Craje C, Krijnen W, Hobbelen H, Van Der Schans C. What type, or combination of exercise can improve preferred gait speed in older adults? A meta-analysis. BMC Geriatr. 2015 Jul 1;15:72. doi: 10.1186/s12877-015-0061-9. PMID 26126532
- [Background] Madeira, J., Silva, C., Marcelino, L., & Ferreira, P. (2015). Assistive Mobile Applications for Dyslexia. Procedia Computer Science, 64, 417-424.
- [Background] Ribeiro J, Souza DN, Costa AP. Qualitative research in the area of health: the whys and wherefores. Cien Saude Colet. 2016 Aug;21(8):2324. doi: 10.1590/1413-81232015218.15612016. No abstract available. English, Portuguese. PMID 27557004
- See also: This link is from the official site of Nursing School of Coimbra, and it refers to MIND&GAIT Project. — https://www.esenfc.pt/pt/page/100004128?idMenu=401
- See also: This link is from the official site of COMPETE2020, and it refers to MIND&GAIT Project. — http://www.poci-compete2020.pt/newsletter/detalhe/Proj23822_MInd&Gait